CLINICAL TRIAL: NCT03603145
Title: Immediate Versus Delayed Insertion of Intrauterine Contraception at the Time of Medical Abortion- An Open-label, Randomized, Multicenter Study
Brief Title: Immediate Versus Delayed Insertion of Intrauterine Contraception After Medical Abortion
Acronym: INTRAM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, Associate professor, senior consultant obstetrics and gynecology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTRAM version III
Record Dates: First submitted 2018-04-25; First posted 2018-07-27 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate insertion (Experimental): Randomized to insertion within 48 hours of medical abortion
  Interventions: Procedure: Immediate insertion
- Standard Insertion (No Intervention): Insertion at 2-4 weeks post medical abortion

INTERVENTIONS:
Procedure: Immediate insertion — Immediate insertion of intrauterine contraception within 48 hours of medical abortion
  Arms: Immediate insertion

SUMMARY:
PICO:

Population:

Women with unwanted pregnancy having a medical abortion and fulfilling inclusion and without exclusion criteria and opting for IUC as post abortion contraception. The medical abortion will be carried out according to the Swedish national evidence based guidelines.

Intervention:

Randomized to insertion of IUC within 48 hours after medical abortion.

Control:

Randomized to insertion of IUC at the time of a follow-up visit scheduled 2 to 4 weeks after the abortion according to routine care.

Objectives:

Evaluation of use of IUC, feasibility, safety, compliance, and acceptability of immediate insertion of IUC 0 to 48 hours after medical abortion compared with delayed IUC insertion at 2 to 4 weeks post abortion. The primary outcome measure will be the use of IUC at 6 months in both groups evaluated by telephone calls/emails follow up.

Time plan: Planning: -March 2018 Study start: May 2018 End of recruitment: April 2020 Last patient Last visit April 2021 Analysis: 2021 Report of primary outcome and Safety: 2021

DETAILED DESCRIPTION:
Today 90 percent of terminations of pregnancy are medical abortions. Approximately 33 000 medical abortions are performed in Sweden each year and 20-30 percent of these women opt for IUC as post abortion contraception. Thus, the results of this study potentially affect at least 6600-9900 women every year in Sweden alone. A disadvantage with medical abortion compared with surgical abortion is the standard practice of delayed insertion of IUC. It has been shown that 42 percent of women scheduled for delayed insertion after surgical abortion did not return for the follow up and IUC insertion.(5) This problem is common also in medical abortion practice. Immediate insertion could lead to insertion rates close to 100 percent. However, this practice has not been studied for medical abortion.

The background for this trial is the belief that a higher rate of insertion of IUC, perhaps close to 100 percent, within 48 hours after medical abortion, can compensate more than well for a potentially higher rate of expulsion at immediate insertion. A clinically significant difference in IUC use at six months following the medical abortion of at least 20 percent is expected.

This large multicenter, randomized, patient centered clinical trial will investigate the effectiveness, feasibility, continued use, safety and acceptability of immediate insertion of intrauterine contraception within 0-48 hours after a completed medical abortion when compared to delayed IUC insertion at 2-4 weeks post abortion which is current practice.

Aim To study use, safety and patient acceptability of intrauterine contraception after immediate insertion compared with standard insertion 2-4 weeks post medical abortion at 3, 6 and 12 months post abortion.

Drug:

Mirena® (LNG-IUS 52mg), Kyleena® (LNG-IUS 19.5mg), Jaydess® (LNG-IUS 13.5 mg), NovaT® (Cu-IUD, medical device, but due to use outside indication it is included in this application)

Design:

Open label, randomized, controlled, multicenter study. Phase III (therapeutic confirming).

Primary objective:

To study if immediate insertion of intrauterine contraception is superior to insertion at 2-4 weeks post abortion with regard to number of women using IUC as contraception at 6 months post abortion.

Variable:

The proportion of women in each group (immediate or delayed) using IUC as contraception at 6 months post abortion (use vs non-use).

Secondary objectives:

To study if immediate insertion of intrauterine contraception is non-inferior to delayed insertion with regard to safety and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* eligible for medical abortion,
* opting for post abortion IUC,
* able and willing to comply with planned follow up.

Exclusion Criteria:

* Contraindication for medical abortion or
* Contraindication for IUC (contraindications may be present for LNG-IUSs but the woman may still choose a Cu-IUD and thereby enter the study),
* inability to give informed consent.
* Septic abortion
* Known hypersensiblity/allergy to levonorgestrel or any of the substances added to the LNG-IUS
* Known abnormal uterine cavity
* Chorioamnionitis
* Abortion associated bleeding > 1000ml
* Uterine atony postabortion
* Placental retention
* Therapeutic antibiotic treatment during abortion, (antibiotics used only as prophylaxis is accepted)
* History of breast cancer
* If any of the following conditions are present an individual evaluation and decision must be done before inclusion: pelvic or genital infection, cervicitis, immunocompromised women, untreated cervical dysplasia, neoplasia in cervix or uterus, acute liver disease or hepatic neoplasia, migraine or other very severe headache, icterus, high uncontrolled blood pressure, serious arterial disease i.e. stroke or myocardial infarction, acute venous thrombosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
use of intrauterine contraception at 6 months post abortion | 6 months post abortion
  use of intrauterine contraception at 6 months post abortion in both groups evaluated through follow up by telephone/email.

SECONDARY OUTCOMES:
Difference in the proportion of women who successfully have the IUC inserted | 10 minutes after (attempted) insertion
  • Difference in the proportion of women who successfully have the IUC inserted (success versus failure),
Expulsion rate following insertion in both groups | 12 months post insertion
  Expulsion rate during 12 months following insertion in both groups evaluated by telephone/email follow up 12 months post abortion (complete, partial or no expulsion.
Continued use of IUC | 12 months post abortion
  • Continued use of IUC at 12 months post insertion evaluated by telephone follow-up (continued use/voluntary discontinued use, involuntary discontinued use including expulsions etc) reasons for discontinuation will be recorded and subsequent use of other contraceptive methods will be noted)
Ease of insertion | 10 minutes after (attempted) insertion
  Ease of insertion according to health care provider (judged as very easy, moderately-, or very difficult)
Pain at time of insertion assessed as millimeters on a 10cm long unmarked Visual Analogue Scale. | 10 minutes after (attempted) insertion
  • pain at time of insertion (women will indicate the pain before insertion, at placement of tenaculum, sound and IUC by putting a vertical mark on a 10 cm long horizontal line with a Visual Analogue Scale (VAS) from 0, indicating no pain to 10 indicating worst imaginable pain. Result will be noted in millimeters and entered into case report forms).
Post-abortion bleeding measured as number of days of fresh bleeding | max 3 months post abortion
  Post-abortion bleeding measured as number of days of uninterrupted fresh bleeding directly following the the abortion.
Post-abortion bleeding measured as number of days of spotting during the first 3 months post abortion | max 3 months post abortion
  Post-abortion bleeding measured as number of days of spotting- excluding fresh bleeding and menstruation- during the first 3 months after the abortion.
Reasons for non-attempted insertion of IUC | within 1 month post abortion
  • Reasons for non-attempted insertion of IUC (change of mind, heavy bleeding, not coming for insertion, staff being unavailable etc),
Complications | 12 months post abortion
  • Complications (adverse events (AE) and serious AE) bleeding requiring any treatment, uterine perforations and cervical tears, infection requiring treatment with antibiotics, hospitalization for any reason, surgical procedures due to heavy bleeding, incomplete abortions, prolonged bleeding or patient request,
Pregnancies occurring during the 12 month follow-up | 12 months post abortion
  • Pregnancies occurring during the 12 month follow-up (planned and unplanned, wanted and unwanted, pregnancy outcomes- ectopic, miscarriage, abortion, molar, kept pregnancy),
proportion of women who would recommend immediate or delayed insertion of IUC post abortion | 12 months post abortion
  • proportion of women who would recommend immediate and delayed insertion of IUC by asking women if they would recommend the procedure to a friend (yes/no, asked at the time of insertion and at the 3, 6 and 12 month follow up),
proportion of women who would recommend IUC for post abortion contraception | 12 months post abortion
  • Proportion of women who would recommend IUC as post abortion to a friend (yes/no) asked at the time of insertion and at the 3, 6 and 12 month follow up),
The proportion of surgical procedures | 3 months post abortion
  • The proportion of surgical procedures in total and for each study site (type of procedure, reasons therefore- infection, retained products of conception, prolonged bleeding etc).

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kopp Kallner, MD, PhD, Principal Investigator — Karolinska Institute, danderyd Hospital
Locations (6):
- Sweden (6):
  - Falun Hospital, Falun
  - Sahlgrenska Hospital, Gothenburg
  - Danderyd Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - South General Hospital, Stockholm
  - Uppsala Academiska Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hogmark S, Envall N, Gemzell-Danielsson K, Kopp Kallner H. One-year follow up of contraceptive use and pregnancy rates after early medical abortion: Secondary outcomes from a randomized controlled trial of immediate post-abortion placement of intrauterine devices. Acta Obstet Gynecol Scand. 2023 Dec;102(12):1694-1702. doi: 10.1111/aogs.14662. Epub 2023 Aug 23. PMID 37614066